CLINICAL TRIAL: NCT03870191
Title: Comparison of Therapeutic Effects of Trigger Point Injection and Twin Nerve Block in Chronic Myofascial Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers University (Other)
Responsible Party: Principal Investigator, Sowmya Ananthan, Principal Investigator, Rutgers University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro20160000530
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Myofascial Pain - Dysfunction Syndrome of TMJ; Trigger Point Pain, Myofascial; Nerve Block
MeSH Terms: conditions — Temporomandibular Joint Disorders; Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Twin Block Group (Active Comparator): This group will receive twin block injections.
  Interventions: Other: Injection of either twin block or trigger point injection.
- Trigger Point Injection Group (Active Comparator): This group will receive trigger point injections.
  Interventions: Other: Injection of either twin block or trigger point injection.

INTERVENTIONS:
Other: Injection of either twin block or trigger point injection. — Study participants will be randomized into either group and will receive the intervention.

SUMMARY:
To see if there is there any difference in the treatment outcomes/results such as changes in pain intensity in patients with myofascial pain who have been treated with trigger point injections or twin block?

DETAILED DESCRIPTION:
Most treatment approaches for chronic myofascial pain are not evidence-based. Studies are usually controversial. Most are short-term, non-randomized. An essential limitation has been the lack of standardization of diagnosis. Some studies do not differentiate between joint pain and muscle pain, which can significantly affect the outcome of the treatment provided.

Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) was recently published and validated. Their protocol allows standardization of the assessment and diagnosis of patients with temporomandibular disorder, including myofascial pain.

To the investigator's knowledge, no previous prospective, randomized study has been conducted demonstrating the treatment outcomes of either trigger point injections or twin block in patients with chronic myofascial pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Myofascial pain with referral based on the DC/TMD criteria
* Pain on the masseter and or temporalis muscles
* Pain present for at least 3 months

Exclusion Criteria:

* Generalized muscle disorder such as fibromyalgia
* Subjects on chronic pain medication
* Subjects who are known to have hypersensitivity to the local anesthetics.
* Pregnant women. A pregnancy test will not be given before subject enrollment. Women of childbearing ages will be asked verbally if they are pregnant. If they are unsure, then they will be excluded from the study.
* Subjects with cognitive problems e.g. Alzheimer's disease.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-06-21 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Pain relief: numerical pain scale | 6 months
  The pain relief received from each injection will be measured using the numerical pain scale. This scale is between 0-10 with 0 meaning no pain and 10 is the most pain.Higher values represent worse pain.

CONTACTS AND LOCATIONS:
Overall Officials: Rafeal Benoliel, BDS, Study Director — Rutgers School of Dental Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ananthan S, Kanti V, Zagury JG, Quek SYP, Benoliel R. The effect of the twin block compared with trigger point injections in patients with masticatory myofascial pain: a pilot study. Oral Surg Oral Med Oral Pathol Oral Radiol. 2020 Mar;129(3):222-228. doi: 10.1016/j.oooo.2019.09.014. Epub 2019 Oct 13. PMID 32009005